CLINICAL TRIAL: NCT06453343
Title: Multicenter Randomized Controlled Trial Comparing Surgical Approaches to the Cochlea for the Slim Modiolar Electrode: Assessing Intracochlear Trauma Using Intraoperative Electrocochleography Measurements and Preservation of Residual Hearing
Brief Title: Clinical Trial to Compare Two Surgical Approaches to the Cochlea
Acronym: BULLS-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: GZA Ziekenhuizen Campus Sint-Augustinus (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL85808.091.23
Record Dates: First submitted 2024-04-29; First posted 2024-06-11 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cochlear Implants; Hearing Loss, Sensorineural
Keywords: Surgical approach; Round Window; Cochleostomy; Electrocochleography; Imaging; Residual hearing preservation
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cochleostomy (Active Comparator): When employing the cochleostomy approach, a carefully positioned opening will be drilled anterior-inferior to the eRW membrane.
  Interventions: Procedure: Surgical approach: cochleostomy or extended round window
- extended Round Window (Active Comparator): In case of the extended round window approach, the scala tympani will be accessed through the extended round window technique, involving the creation of a round window margin cochleostomy.
  Interventions: Procedure: Surgical approach: cochleostomy or extended round window

INTERVENTIONS:
Procedure: Surgical approach: cochleostomy or extended round window — Surgical placement of a cochlear implant electrode array

SUMMARY:
This is a prospective multicenter multinational randomized control trial. The duration of the study for the individual patient will be approximately 1 year (pre-operative assessments, 1 week, 3 months and 12 months follow-up assessments). Participants will be randomized to one of two surgical approaches: eRW or CO, with a 1:1 allocation in a parallel design.

DETAILED DESCRIPTION:
Rationale: Preserving residual hearing in cochlear implant (CI) surgery has gained significant attention. It not only signifies minimally invasive implantation but also supports natural sound perception and enables electrical-acoustic stimulation, enhancing sound localization, music appreciation, and speech recognition in noisy environments. Using the Cochlear™ Nucleus® CI with Slim Modiolar electrode (Cochlear Ltd., Sydney, Australia), potential sites of residual hearing loss in surgery include approaches to the cochlear lumen, potential damage during entry, and damage during electrode insertion. Studies comparing different surgical approaches (cochleostomy (CO) and extended round window (eRW)) show varied results. Electrocochleography (ECochG) can be used to indicate intracochlear damage during electrode insertion, however, the variability observed in ECochG responses during cochlear implantation remains significant. Moreover, ECochG has not yet been used to monitor cochlear functions throughout every phase of surgery, including the insertion of the sheath or stabilization of the electrode lead.

Objective: The aim of this study is to investigate whether the type of surgical approach to the cochlea; CO or eRW using the CI632 affects the final residual hearing and secondarily, intracochlear trauma and electrode position, as determined by pure tone audiometry, EcochG and imaging.

Study population: Adult CI candidates with post-lingual onset of severe to profound hearing loss, who are scheduled to receive a Nucleus CI632 with a slim modiolar electrode array and have a preoperative audiometric low-frequency average air conduction threshold of <80 decibel (dB) hearing level at 500 Hz in the ear to be implanted.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and older who have clinically established post-linguistic sensorineural hearing loss.
* CI candidate based on local or national reimbursement criteria.
* Cochlear implantation with a CI632.
* Preoperative 500 Hz pure-tone air conduction threshold <80 dB hearing level (HL) in the ear to be implanted.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Previous or existing CI recipient.
* Ossification or other anatomical abnormalities of the cochlea or its windows possibly affecting normal electrode array insertion.
* Abnormal cochlear nerve anatomy on preoperative CT or MRI.
* Subjects who are unable to undergo CT or MRI.
* Deafness due to acoustic nerve or central auditory pathway lesions.
* Diagnosis of auditory neuropathy.
* Active middle ear infection.
* Additional handicaps that would prevent participation in study evaluations.
* Unrealistic expectations from the participant regarding the possible benefits, risks, and limitations inherent to the CI procedure and the investigation.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Residual hearing | 3-months postoperatively
  The difference in residual hearing per group (eRW or CO) between pre- and postoperative pure tone thresholds, averaged at 500, 750 and 1000 Hz (PTAlow).

SECONDARY OUTCOMES:
ECochG thresholds after multiple surgery stages | Intraoperatively
  ECochG thresholds with a promontory recording electrode after the following surgery stages: a) posterior tympanotomy (baseline), b) drilling for RW membrane exposure, c) completion of the approach to implantation (CO or eRW), d) sheath insertion, e) electrode array insertion, f) sheath withdrawal, and g) positioning of the electrode lead.
Intracochlear electrode position | 3-months postoperatively
  The position of electrode contacts relative to the modiolus and the angular insertion depth (AID), as assessed with pre- and post-operative CT-scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No